CLINICAL TRIAL: NCT00000702
Title: A Multicenter Placebo-Controlled Double-Blind Trial to Evaluate Azidothymidine (AZT) Treatment of the AIDS Dementia Complex and Central Nervous System (CNS) Human Immunodeficiency Virus (HIV) Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 005; 10981 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: AIDS Dementia Complex; HIV Infections
Keywords: AIDS Dementia Complex; Zidovudine
MeSH Terms: conditions — AIDS Dementia Complex; HIV Infections | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To test whether zidovudine (AZT) is useful as a treatment for the neurologic syndrome called AIDS dementia complex. To determine how long AZT takes to reach cerebral spinal fluid (CSF), how long, and at what concentration it is found there.

HIV infection can result in impairment in the function of the brain and spinal cord, leading to disturbances in the ability to think clearly and in strength and coordination. This disorder, which has been called the AIDS dementia complex, may be due to a direct effect of HIV on the nervous system. It is known that AZT does get into the brain to some extent, where it may reduce growth of HIV. It is hoped that AZT will stabilize or improve the symptoms of the AIDS dementia complex.

DETAILED DESCRIPTION:
HIV infection can result in impairment in the function of the brain and spinal cord, leading to disturbances in the ability to think clearly and in strength and coordination. This disorder, which has been called the AIDS dementia complex, may be due to a direct effect of HIV on the nervous system. It is known that AZT does get into the brain to some extent, where it may reduce growth of HIV. It is hoped that AZT will stabilize or improve the symptoms of the AIDS dementia complex.

The study is done in 2 stages. In Stage 1, patients are randomized to receive placebo or 1 of 2 doses of AZT. Stage 1 lasts for 4 months. In Stage 2, patients who were initially treated with placebo are randomized again and all patients receive AZT. Stage 2 lasts an additional 12 months, during which time there are periodic medical and neurologic evaluations. Before beginning treatment, all patients have a lumbar puncture and a computerized tomographic (CT) scan of the brain. The lumbar puncture is repeated twice during and once at the end of Stage 1; the CT scan is also repeated at the end of Stage 1. Patients receiving AZT in either stage 1 or Stage 2 are seen by their physicians every week for the first 4 weeks and every other week thereafter for the first 4 months of receiving the drug. After 4 months, patients are seen by their physicians at 4 to 12 week intervals.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aspirin, in modest doses.
* Ibuprofen, in modest doses.
* Maintenance antibiotic therapy posttherapy for an AIDS-defining opportunistic infection.

Concurrent Treatment:

Allowed:

* Blood transfusion if cardiovascular status is compromised.

Exclusion Criteria

* Active substance abuse.

Co-existing Condition:

Patients with the following conditions will be excluded:

* Concurrent or previous central nervous system infections or neoplasms.
* Active AIDS-defining opportunistic infection.
* Severe premorbid psychiatric illness.
* Confounding neurological disease.
* Concurrent neoplasms.

Concurrent Medication:

Excluded:

* Maintenance methadone or naltrexone.
* Acetaminophen.
* Mood- or central nervous system-altering drugs.
* Zidovudine for Pneumocystis carinii pneumonia (PCP).
* Acyclovir.
* Rifampin or derivatives.
* Drugs with antiretroviral activity.
* Experimental agents.

The following patients will be excluded from the study:

* Patients requiring ongoing therapy for an AIDS-defining opportunistic infection.
* Patients with a history of Mycobacterium avium intracellulare infection.
* Patients with a history of Pneumocystis carinii pneumonia infection.
* Patients with a daily temperature of 38 degrees C or more for 1 month.

Prior Medication:

Excluded:

* Zidovudine (AZT).
* Excluded within 14 days of study entry:
* Systemic anti-infectives.
* Excluded within 30 days of study entry:
* Immunomodulators and biologic response modifiers.
* Any investigational agent.
* Cytotoxic chemotherapy for Kaposi's sarcoma.

Prior Treatment:

Excluded:

* Radiation therapy.

Patients must demonstrate the following clinical and laboratory findings:

* No currently active AIDS-defining opportunistic infections.
* One negative blood culture for Mycobacterium avium intracellulare within 4-6 weeks prior to study entry.
* Constitutionally well without persistent fever.
* Less than 25 Kaposi's sarcoma lesions and less than 10 new lesions during the 30 days prior to study entry. Patients may have stable or indolently progressive mucocutaneous Kaposi's sarcoma.
* Characteristic clinical symptoms and signs of AIDS dementia complex.
* Abnormalities on 2 or more of 7 neuropsychological motor tests in the Neurological Screening Battery.
* Estimated premorbid IQ equal to or greater than 70 (+ or - 5), which is consistent with completion of sixth grade.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 315
Dates: Study Completion 1990-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R Price, Study Chair
Locations (21):
- United States (21):
  - UCLA CARE Ctr, Los Angeles, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Stanford Univ School of Medicine, Stanford, California
  - Univ of Miami School of Medicine, Miami, Florida
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Louisiana State Univ Med Ctr / Tulane Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Beth Israel Med Ctr / Peter Krueger Clinic, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Sidtis JJ, Gatsonis C, Price RW, Singer EJ, Collier AC, Richman DD, Hirsch MS, Schaerf FW, Fischl MA, Kieburtz K, et al. Zidovudine treatment of the AIDS dementia complex: results of a placebo-controlled trial. AIDS Clinical Trials Group. Ann Neurol. 1993 Apr;33(4):343-9. doi: 10.1002/ana.410330403. PMID 8489204
- [Background] Price RW, Koch MA, Sidtis JJ, Feinberg J, Collier A, Kennedy C, Singer E, Price S. Zidovudine (AZT) treatment of the AIDS dementia complex (ADC): results of a placebo-controlled, multicentered therapeutic trial. Int Conf AIDS. 1989 Jun 4-9;5:407 (abstract no WBP331)